CLINICAL TRIAL: NCT02046109
Title: Replacement Versus Repair of Composite Restorations, a Randomized Controlled Trial
Brief Title: Study of the Success and Survival of Dental Composite Restorations Being Repaired Instead of Being Replaced
Acronym: RVR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of logistic problems, we could not recruit any patient.
Sponsor: Dalhousie University (Other)
Responsible Party: Principal Investigator, Pierre-Luc Michaud, Assistant Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DalDent-2014-01
Record Dates: First submitted 2014-01-23; First posted 2014-01-27 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Failing Dental Composite Restorations
Keywords: Repair; Replace; Composite; restoration; failing dental restoration; filling; dental; dentistry
MeSH Terms: interventions — Wound Healing; Filtek Supreme

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Repair (Experimental): Subjects in the Repair group will be given a local anesthetic only if required (i.e. for restorations extending gingivally or on exposed dentin surface) as per usual clinical protocol. The existing restoration will not be removed. The surface of the existing restoration will be roughened with a Brasseler 8856 bur without extending to the surrounding enamel (except is the defect being repaired is adjacent to enamel). No accessory groves/pits for retention will be prepared. To repair the restoration, the surface will be etched using 35% phosphoric acid, and then 3M ESPE Scotchbond Universal Adhesive System followed by 3M ESPE Filtek Supreme Ultra Universal Restorative composite will be used as per the manufacturer's instructions.
  Interventions: Procedure: Repair
- Replace (Active Comparator): Subjects in the Replace group will be given local anesthetic (an injection of 2% lidocaine with 1:100 000 epinephrine). The type of injection and dosage of anesthetics will be dependent on the tooth being treated, and will follow the usual protocol used in the Dalhousie Dentistry undergraduate clinics. The existing composite restoration will then be removed and the peripheral enamel beveled if not already beveled. To restore the tooth, the surface will be etched using 35% phosphoric acid, and then 3M ESPE Scotchbond Universal Adhesive System followed by 3M ESPE Filtek Supreme Ultra Universal Restorative composite will be used as per the manufacturer's instructions.
  Interventions: Procedure: Replace

INTERVENTIONS:
Procedure: Repair
  Other Names: Scotchbond Universal; Filtek Supreme
  Arms: Repair
Procedure: Replace
  Other Names: Scotchbond Universal; Filtek Supreme
  Arms: Replace

SUMMARY:
The objective of this trial is to compare the success (as assessed by a pre-defined set of outcome) of failing composite resin restorations that are repaired using diamond bur induced surface abrasion, to those that are completely replaced.

It is hypothesized that both treatment will have comparable success rate.

DETAILED DESCRIPTION:
This study is a single-blind randomized non-inferiority trial using parallel groups.

Patients recruited into the study will be randomly assigned to one of two treatment groups. Subjects allocated to Group 1 will have their defective restoration completely replaced while subjects allocated to Group 2 will have their defective restoration repaired.

The success of the treatments will be assessed immediately following the intervention (baseline) and 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the Dalhousie University Dental Clinic who are:
* Age 18 and over
* Capable of providing informed consent
* Asymptomatic permanent teeth with class III, IV, V or veneer composite restorations on the facial/buccal surface, requiring treatment (e.g. stain, chipping or color discrepancy).
* Restoration must present with a portion (mesial, distal, gingival or occlusal) that can be completely retained to allow repair.

Exclusion Criteria:

* Patients with contra-indications for regular dental treatment based on their medical history
* Teeth with active caries
* Teeth with multiple overlapping composite restorations
* Patients with uncontrolled periodontal disease
* Restorations smaller than 3mm diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Success rate | 12-month
  The primary outcome will be the success of the restoration. This will be assessed using the modified U.S. Public Health Service (USPHS) criteria as first described by Cvar and Ryge (1971) and adapted by Wilson et al (2002).

SECONDARY OUTCOMES:
Survival | 12-month

CONTACTS AND LOCATIONS:
Locations (1):
- Dalhousie University Faculty of Dentistry, Halifax, Nova Scotia, Canada

REFERENCES:
- See also: Dalhousie University Faculty of Dentistry Web Site — http://www.dal.ca/faculty/dentistry.html